CLINICAL TRIAL: NCT05325554
Title: Research on Multi-mode Rehabilitation of Abdominal Tumor Patients With Simultaneous Radiotherapy and Chemotherapy Based on Mobile Medicine.
Brief Title: Multi-mode Rehabilitation of Abdominal Tumor Patients Undergoing Concurrent Chemoradiotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Zhou Fuxiang, Clinical Professor of Zhongnan Hospital, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCCSC AB05
Record Dates: First submitted 2022-03-08; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Concurrent Chemoradiotherapy;Nutrition；Multimodal Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research Group (Experimental): multi-mode rehabilitation
  Interventions: Behavioral: Multimodal rehabilitation
- control group (No Intervention): control group

INTERVENTIONS:
Behavioral: Multimodal rehabilitation — Multimodal rehabilitation
  Arms: Research Group

SUMMARY:
The investigators carry out a multi center, randomized controlled clinical study to analyze the impact of the whole process multi-mode rehabilitation management (nutrition-Sports-Psychology) on the nutritional status, physical status, psychological status, treatment side effects and the completion rate of radiotherapy and chemotherapy of patients with abdominal tumors; To explore and establish a multi-mode rehabilitation management path for patients with malignant tumors undergoing concurrent radiotherapy and chemotherapy.

DETAILED DESCRIPTION:
Research shows that the combination of early nutritional intervention and psychological palliative intervention can improve the quality of life of patients, reduce the probability of depression, improve the prognosis of patients and prolong the overall survival time for up to two months. The research of Peking University Cancer Hospital in China shows that early nutrition and psychological palliative intervention can improve the prognosis of patients with advanced esophageal cancer and prolong the overall survival by nearly three months. The first mock exam (including exercise, nutrition and Psychology) seems to be more effective than a single model of pre rehabilitation. Therefore, the current triple rehabilitation strategy is advocated, namely, high intensity aerobic exercise during the waiting period, nutritional support based on protein supplementation, and psychological support to eliminate anxiety. Tumor multimodal rehabilitation has received more and more attention, but there is no clinical research on the "triple multimodal rehabilitation" of nutrition + Exercise + psychology in patients with abdominal tumor concurrent radiotherapy and chemotherapy. Therefore, the research on the impact of whole process multimodal rehabilitation (nutrition-Exercise-Psychology) on patients with abdominal tumor concurrent radiotherapy and chemotherapy has been carried out, It has important scientific significance and value to promote the rehabilitation and development of tumor patients undergoing concurrent radiotherapy and chemotherapy.

In this study,the investigators carry out a multi center, randomized controlled clinical study to analyze the impact of the whole process multi-mode rehabilitation management (nutrition-Sports- Psychology) on the nutritional status, physical status, psychological status, treatment side effects and the completion rate of radiotherapy and chemotherapy of patients with abdominal tumors; To explore and establish a multi-mode rehabilitation management path for patients with malignant tumors undergoing concurrent radiotherapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed as abdominal malignant tumor by pathology and / or cytology and intend to receive concurrent radiotherapy and chemotherapy;
2. Estimated survival time ≥ 3 months;
3. ECoG score 0-1;
4. The physical activity is acceptable, and the human body composition analysis and 6-minute walking test can be carried out;
5. Have reading comprehension ability and be able to complete the questionnaire.

Exclusion Criteria:

1. Clinically significant cardiovascular diseases, such as heart failure (NYHA grade III-IV), uncontrolled coronary heart disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension or history of myocardial infarction in the past 1 year;
2. Neurological or psychiatric abnormalities affecting cognitive ability, including central nervous system metastasis;
3. uncontrolled systemic diseases, such as poorly controlled diabetes mellitus;
4. Allergic to milk, whey protein, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Completion rate of concurrent chemoradiotherapy | up to 12 weeks
  Completion rate of concurrent chemoradiotherapy
Changes in grip strength | up to 12 weeks
  Changes in grip strength
Improvement of nutritional status | up to 12 weeks
  PG-SGA score

SECONDARY OUTCOMES:
Side effects of concurrent radiotherapy and chemotherapy | up to 12 weeks
  Side effects of concurrent radiotherapy and chemotherapy
disease free survival | up to 12 weeks
  disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hopital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No